CLINICAL TRIAL: NCT04187326
Title: Feed Forward Visual System Function In High Trait Anxiety
Brief Title: Assessing Visual Processing in High Anxiety
Acronym: ALPHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Elliot Kale Edmiston, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19010289; 1K01MH117290-01A1 (NIH)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Anxiety
Keywords: visual processing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study team will use a waitlist-control design. A subset of participants will return to complete visual training using the Micro Expression Training Tool (METT). Half of these participants will complete the task at their first follow up visit (approximately six months post scan), and half will complete the task at their second follow up visit (approximately twelve months post scan).
  The METT presents videos of micro expressions; participants receive real-time feedback following forced choice emotional identification. The METT includes a brief pre-test, training, and then a post-test. We will collect performance accuracy data. This behavioral task will provide preliminary feasibility data for the development of interventions with visual system targets by helping the investigators determine if the METT is tolerable in individuals with high trait anxiety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6 Month Micro Expression Training Task (Experimental): The Micro Expression Training Task (METT) presents videos of subtle emotional face expressions; participants receive real-time feedback following forced choice emotional identification. The METT includes a brief pre-test, training, and then a post-test.
  Interventions: Behavioral: Facial Microexpression Training
- 12 Month Micro Expression Training Task (Experimental): The Micro Expression Training Task (METT) presents videos of subtle emotional face expressions; participants receive real-time feedback following forced choice emotional identification. The METT includes a brief pre-test, training, and then a post-test. Participants in this group will complete this task twelve month after their first visit.
  Interventions: Behavioral: Facial Microexpression Training

INTERVENTIONS:
Behavioral: Facial Microexpression Training — The METT is a well-validated task designed to improve perception of subtle changes in facial expressions, termed microexpressions. Participants with high trait anxiety will return to the lab approximately six months post scan visit to complete this computer-based task. They will receive feedback during the task on their accuracy.

SUMMARY:
High trait anxiety, a stable personality trait, is a risk factor for psychiatric disorders. Individuals with high trait anxiety have difficulty differentiating safety from threat, including visual information like emotional faces. This study aims to characterize visual system function in high trait anxiety. A portion of this study involves an intervention. For the intervention portion, a subset of participants will be asked to return for a lab visit upon completing the first portion of the study (multimodal magnetic resonance imaging (MRI) scan). During this follow up visit, participants will complete a computer task that involves looking at faces and identifying emotions. Participants will complete this task either six months or twelve months after their MRI scan visit. Results from this research have the potential to inform novel therapies that target the visual system in individuals at risk for the development of psychiatric disorders.

DETAILED DESCRIPTION:
The purpose of this study is to understand how people with anxious personalities process emotional facial expressions. The intervention portion of this study is part of a larger study. The first portion of this study consists of a screening visit with questionnaires, and a second visit with a magnetic resonance imaging (MRI) scan and short computer tasks.

For the intervention portion of this study, a subset of participants will return to the lab for an in-person visit either six or twelve months after their MRI scan. This visit will last approximately two hours. Participants will be asked to complete a computer task where they will be asked to identify emotional face expressions and receive feedback on their performance. They will also complete questionnaires about their mood and emotions.

The primary purpose of this research is to gather scientific information about how people with anxiety process social and emotional information.

ELIGIBILITY:
Inclusion Criteria:

* Young adults varying continuously in trait anxiety as assessed by the Spielberger State Trait Anxiety Inventory (STAI).
* HTA participants with STAI trait scores of ≥44

Exclusion Criteria:

* contraindication to MRI
* history of head trauma or loss of consciousness
* major medical or neurological illness
* current psychiatric medication usage or use in the last three months
* alcohol/substance abuse or dependence and/or illicit substance use (excepting cannabis) in the last three months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot K Edmiston, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Massachusetts Chan School of Medicine, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants complete baseline visit and functional MRI scan prior to randomization to trial arms. Only participants with high trait anxiety, as assessed by the Spielberger Trait Anxiety Inventory at baseline visit, are randomized to a trial arm.
Period: Overall Study
Arm/Group | 6 Month Micro Expression Training Task | 12 Month Micro Expression Training Task
Started | 7 | 8
Completed | 5 | 6
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Computer error- task was only partially completed. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 Month Micro Expression Training Task | 12 Month Micro Expression Training Task | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.08 (3.05) | 22.91 (3.29) | 23.92 (3.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of the Micro Expression Training Task in Individuals With High Anxiety
Description: Rates of completion of the behavioral task
Time Frame: six or twelve months post-scan visit
Population: Participants from a larger study with high trait anxiety were randomized to either a 6 month or 12 month arm.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 Month Micro Expression Training Task | 12 Month Micro Expression Training Task
Number analyzed (Participants) | 7 | 8
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: 1 year
Description: AE definition is the same as clinicaltrials.gov definitions
Arm/Group | 6 Month Micro Expression Training Task | 12 Month Micro Expression Training Task
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT04187326/Prot_001.pdf
  • Informed Consent Form (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT04187326/ICF_002.pdf